CLINICAL TRIAL: NCT01990716
Title: Quantitative Analysis of Lipid Mediators in Colonic Biopsies From Patients With Inflammatory Bowel Diseases and From Control Patients.
Brief Title: Lipid Mediators in Colonic Biopsies as Biomarkers of Disease Activity of Inflammatory Bowel Diseases
Acronym: MICILIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12 393 02; AOL 2012 (Other: University of Toulouse)
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease
Keywords: Adult; Colonoscopy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBD patients (Other): Patients (diagnosed with IBD) having a screening colonic biopsy
  Interventions: Other: Colonic Biopsy
- Control Group (Other): individuals undergoing screening colonic biopsy for colon cancer or polyp detection, who have not been diagnosed with any intestinal pathology.
  Interventions: Other: Colonic Biopsy

INTERVENTIONS:
Other: Colonic Biopsy — Colonoscopy or coloscopy can provide a visual diagnosis and grants the opportunity for biopsy or removal of suspected colorectal cancer lesions.
  The endoscope is then passed through the anus up the rectum, the colon, and ultimately the terminal ileum. The endoscope has a movable tip and multiple channels for instrumentation, air, suction and light. Biopsies are frequently taken for histology, needed for cancer or IBD diagnosis.
  Extra-biopsies for research purpose will only be performed if the clinician decides that they are necessary for the clinical diagnosis or for the disease follow-up.
  For this protocol, collecting these extra biopsies should last under 5 minutes and should not extend the procedure by more than this time.

SUMMARY:
We will quantify one of the lipid compounds (5,6 epoxy eicosatrienoic acid (5,6 EET), 5,6- EpoxyEicosaTrienoic acid) in colonic biopsies of Inflammatory Bowel Disease patients. We will evaluate its possible use as a pathological activity biomarker and its potential as a therapeutic target.

We hypothesized that 5,6-EET is present in human colonic tissues in varying quantities depending on the pathological state of the IBD patient.

DETAILED DESCRIPTION:
The project is an exploratory physiopathological/translational pilot study, aiming at understanding the relative importance of the lipid compounds, especially 5,6-EET, in Inflammatory Bowel Diseases.

Using mass spectrometry, 5,6-EET and other 33 lipid metabolites will be quantified in situ in colonic biopsies from IBD patients and from control patients. We will compare quantities of 5,6-EET in inflammatory and non-inflammatory zones of biopsies from IBD patient to biopsies from control patient. We will establish a cluster of lipid compounds associated with pathological activity. We will determine the exposed profile of receptor lipid mediators expressing to the 5,6-EET lipid compound and one of its signalization.

All data will be submit to statistical analysis to confirm relevance.

We expect this pilot study to help us define 5,6-EET and other components of the same metabolic family as markers for IBD activity. It could point lipid mediators and their receptors as potential new therapeutic targets.

It will increase our knowledge on current treatment efficiency by evidencing lipid markers for the inflammatory condition.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA FOR IBD PATIENTS

* Major/18 years and older
* Covered by a health insurance plan
* Patient having a screening colonoscopy for/with a suspicion of IBD or, IBD Patient, either in acute phase or in remission, having a therapeutic colonoscopy as part of his/her regular follow- up/usual care
* Must be able to understand and voluntarily sign an informed consent prior to any study procedures

INCLUSION CRITERIA FOR IBD PATIENTS

* Major/18 years and older Covered by a health insurance plan
* Patients having a screening colonoscopy for polyp or cancer detection or patient undergoing a colic resection
* Must be able to understand and voluntarily sign an informed consent prior to any study procedures

Exclusion Criteria:

EXCLUSION CRITERIA FOR IBD PATIENTS

* Unable to comprehend the full nature and purpose of the study, and/or difficulty in communicating with the investigator
* Deprivation of liberty by administrative or legal decision
* Any other pathological or psychological condition considered by the investigator as interfering with the study (pregnancy, breastfeeding, cancer detection, AIDS, celiac disease)
* Participation in another biomedical research/clinical trial with experimental medication within the last 3 months prior to the selection visit or patients still within a biomedical research exclusion period
* Presence of cancerous lesions
* Anatomopathological results excluding the possibility of an IBD
* Contra-indications to carrying out a lower digestive endoscopy

EXCLUSION CRITERIA FOR CONTROL PATIENTS

* Unable to comprehend the full nature and purpose of the study,
* and/or difficulty in communicating with the investigator
* Deprivation of liberty by administrative or legal decision
* Participation in another biomedical research/clinical trial with experimental medication within the last 3 months prior to the selection visit or patients still within a biomedical research exclusion period
* Contra-indications to carrying out a lower digestive endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Measure of 5,6-EET quantity in a colonic biopsy | 5 minutes
  Mass spectrography analysis of the biopsies will be performed each time at least 10 samples are available

SECONDARY OUTCOMES:
Nature and quantity of Lipid metabolites as a function of the patient clinical profile (mapping) | 5 minutes
  This measure will be performed at the same time than the first outcome measure (each time at least 10 samples are available).

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Alric, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rahabi M, Jacquemin G, Prat M, Meunier E, AlaEddine M, Bertrand B, Lefevre L, Benmoussa K, Batigne P, Aubouy A, Auwerx J, Kirzin S, Bonnet D, Danjoux M, Pipy B, Alric L, Authier H, Coste A. Divergent Roles for Macrophage C-type Lectin Receptors, Dectin-1 and Mannose Receptors, in the Intestinal Inflammatory Response. Cell Rep. 2020 Mar 31;30(13):4386-4398.e5. doi: 10.1016/j.celrep.2020.03.018. PMID 32234475